CLINICAL TRIAL: NCT01569945
Title: Hormonal Stimulation in IUI Treatment: Is Clomifen Combined With Ethinyl Estradiol Better, Worse or Equal to Menopur
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Thomas D'Hooghe, Profsessor Medical Doctor, University Hospital, Gasthuisberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML2436 - 1
Record Dates: First submitted 2012-03-28; First posted 2012-04-03 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Subfertility
MeSH Terms: conditions — Infertility | interventions — Clomiphene; Ethinyl Estradiol; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tablets (Active Comparator): Clomifen (5 days) followed by Ethinyl Estradiol (5 days)
  Interventions: Drug: Clomifen, Ethinyl Estradiol
- human menopausal gonadotropins (Active Comparator): Daily Injections
  Interventions: Drug: Menotropins

INTERVENTIONS:
Drug: Clomifen, Ethinyl Estradiol — starting on day 2 or 3 of the cycle: 1 tablet of Clomifen each day, for 5 days in a row. Dose 50mg or in subsequent cycles, 25 mg or 100 mg or 150 mg. After the 5 days of Clomifen, one tablet of Ethinyl Estradiol 50 mg per day, for 5 days in a row or until beta hCG is injected
  Arms: Tablets
Drug: Menotropins — Starting on day 2 or 3 of the cycle, a daily subcutaneous injection of 37.5 IU or 75.0 IU
  Arms: human menopausal gonadotropins

SUMMARY:
What is the best medication for hormonal stimulation in cycles with high intra-uterine insemination: tablets of Clomifen (5 days) followed by tablets of Ethinyl Estradiol (5 days) or daily injections with Human Menopausal Gonadotropin (Menopur)?

ELIGIBILITY:
Inclusion Criteria:

* women younger than 42 years old
* infertility of at least one year
* normal tubal, pelvic and uterine anatomy
* semen with total motility count of at least 5 million (at least one sample)

Exclusion Criteria:

* premature ovarian failure
* medical history of tubal or ovarian surgery
* tubal or pelvic adhesions

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 371 (Actual)
Dates: Start 2004-09; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | on average 30 days if not pregnant and 12 weeks if pregnant

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D'Hooghe, MD PhD, Principal Investigator — University Hospital, Gasthuisberg
Locations (1):
- Leuven University Fertility Center, Leuven, Vlaams Brabant, Belgium

REFERENCES:
- [Derived] Peeraer K, Debrock S, De Loecker P, Tomassetti C, Laenen A, Welkenhuysen M, Meeuwis L, Pelckmans S, Mol BW, Spiessens C, De Neubourg D, D'Hooghe TM. Low-dose human menopausal gonadotrophin versus clomiphene citrate in subfertile couples treated with intrauterine insemination: a randomized controlled trial. Hum Reprod. 2015 May;30(5):1079-88. doi: 10.1093/humrep/dev062. Epub 2015 Mar 18. PMID 25788569